CLINICAL TRIAL: NCT03858348
Title: A Retrospective rEal-life daTa Study to Assess the Incidence of exaceRbations and Change in Lung functIon Forced Expiratory Volume (FEV1) in Chronic Obstructive Pulmonary Disease ( COPD ) patiEnts receiVing Fluticasone/Salmeterol Fixed Dose Combination (FDC) Comparing to Those Εscalating in Open-triple Fluticasone/Salmeterol, Long Acting Muscarinic Antagonist (LAMA) Combination
Brief Title: A Retrospective rEal-life daTa Study to Assess the exaceRbations and Lung functIon in Chronic Obstructive Pulmonary Disease ( COPD ) patiEnts receiVing Fluticasone/Salmeterol Comparing to Those Εscalating in Open-triple Fluticasone/Salmeterol, Long Acting Muscarinic Antagonist (LAMA) Combination
Acronym: RETRIEVE
Status: Completed | Type: Observational
Sponsor: Elpen Pharmaceutical Co. Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2019-FLSAL-EL-94
Record Dates: First submitted 2019-02-20; First posted 2019-02-28 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: COPD; COPD Exacerbation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- fluticasone / salmeterol treatment: The evaluation of pulmonary function in patients with COPD receiving and maintaining a stable combination of fluticasone / salmeterol (Group A)
- fluticasone / salmeterol and extra LAMA: The evaluation of pulmonary function in patients with COPD receiving and maintaining a stable combination of fluticasone / salmeterol and extra a long-acting muscarinic receptor antagonist (anticholinergic, LAMA) (Group B).

SUMMARY:
Inhaled corticosteroid (ICS)/long-acting β2-agonist (LABA) combination is commonly prescribed to treat COPD; we will perform a retrospective analysis on the effect of adding a long-acting muscarinic receptor antagonist (LAMA) to ICS/LABA combination in COPD.

DETAILED DESCRIPTION:
According to the current guidelines for the treatment of COPD, it is recommended to use combination therapies with different or complementary mechanisms of action . Data suggest that open triple therapy incorporating LAMA with ICS / LABA combination products administered through different delivery devices may be beneficial for improving pulmonary function in patients with COPD. However, there is little evidence of the effect of triple therapy on pulmonary function and the incidence of exacerbations in COPD patients.

ELIGIBILITY:
Inclusion

* Patients with COPD who started treatment with a fixed combination of fluticasone / salmeterol via the Elpenhaler® device after 01/01/2012 and were treated continuously for at least 1 year during the recording period.
* Patients for whom spirometric data are available per monitoring year during recording.
* Patients for whom exacerbation data are available per monitoring year during recording.

Exclusion

•Patients with asthma

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD patients
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
FEV1 | 36 months
  The rate of FEV1 change in patients in both groups A and B during the recording period.
Exacerbations | 36 months
  The number of exacerbations per year of patients in both groups A and B during the recording period.

CONTACTS AND LOCATIONS:
Locations (1):
- Papanikolaou Hospital of Thessaloniki, Thessaloniki, Greece

REFERENCES:
- See also: A retrospective evaluation of lung function and exacerbations in COPD patients-RETRIEVE study European Respiratory Journal 2021 58: PA2402; DOI: 10.1183/13993003. — https://erj.ersjournals.com/content/58/suppl_65/PA2402
- See also: Factors influencing LAMA addition to COPD patients receiving ICS/LABA in clinical practice-RETRIEVE study European Respiratory Journal 2021 58: PA795; DO — https://erj.ersjournals.com/content/58/suppl_65/PA795